CLINICAL TRIAL: NCT06384274
Title: The Effect of Emotional Freedom Technique and Virtual Reality Glasses on Anxiety and Vital Signs in Individuals Receiving Hyperbaric Oxygen Therapy: Randomized Controlled Trials
Brief Title: The Effect of Emotional Freedom Technique and Virtual Reality Glasses on Anxiety and Vital Signs
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Necmettin Erbakan University (Other)
Responsible Party: Principal Investigator, Gülsüm Gürsoy Açıkgöz, Principal Investigator, Necmettin Erbakan University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: NEUniversity
Record Dates: First submitted 2024-04-06; First posted 2024-04-25 (Actual); Last update posted 2024-04-25 (Actual); Status verified 2024-04

CONDITIONS: Anxiety
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Emotional Freedom Technique Group (Experimental): When the patient, who was determined to be in the emotional liberation group, was admitted to the unit, the patient's consent was first obtained; In the first 10 minutes, the patient will fill out the Patient Introduction Form, State Anxiety Scale, Subjective Disturbance Unit Scale and Vital Signs Form in the Unit.
  Emotional liberation technique will be applied and then the subjective disturbance unit score will be recorded. Then the patient will fill out the State Anxiety Scale and Vital Signs Forms and the patient will be informed about the treatment. He will then be taken into treatment. When the patient leaves the treatment, the process will be completed by filling out the State Anxiety Scale, Subjective Disturbance Unit Scale and Vital Signs Form again within 10 minutes.
  Interventions: Other: Emotional Freedom Technique
- Virtual Reality Glasses Group (Experimental): Consent was first obtained for admission differences to the patient unit, which was noted to have virtual reality limits; Patient Introduction Form, State Anxiety Scale, Subjective Disturbance Unit Scale and Vital Tests Form will be filled in the unit.
  Then the virtual reality of life will be explained and glasses will be purchased. Forest/beach/sea video images can be watched in virtual reality. The video is planned to last approximately 10 minutes. The application is planned to take 20-25 minutes. Before the session, the State Anxiety Scale, SUBJECTIVE DISORDER UNIT SCALE and Vital Tests Form will be filled in again, the patient will be informed and then the treatment will be administered.
  Once the treatment is completed, the patient will take a third measurement within 10 minutes and the State Anxiety Scale, Subjective Disturbance Unit Scale and Life Parameters Form will be filled out again.
  Interventions: Other: Virtual Reality Glasses
- Control Group (No Intervention): When the patient determined to be in the control group is admitted to the unit, patient consent was obtained within the first 10 minutes and the Patient Introduction Form, State Anxiety Scale, Subjective Disturbance Unit Scale and Vital Signs Form will be filled in the unit. The patient will be prepared for the treatment, will be given special clothing for the treatment, and will be given standard training for the treatment. Then, the second measurement will be taken just before the patient enters the session. There will be at least 20 minutes between the second measurement and the first measurement. The State Anxiety Scale, Subjective Disturbance Unit Scale and Vital Signs Form will be filled out again. After the treatment process is completed, the patient will be measured for the third time and the process will be completed by filling out the State Anxiety Scale, Subjective Disturbance Unit Scale and Vital Signs Form again.

INTERVENTIONS:
Other: Emotional Freedom Technique — All people have an energy body. If the energy flow is interrupted, emotions such as stress and fear arise. By clicking on energy points to improve energy flow, the individual gets rid of energy blockages.
  Arms: Emotional Freedom Technique Group
Other: Virtual Reality Glasses — It is aimed to reduce the patient's anxiety by making her feel like she7 he is there by watching and listening to relaxing content of the beach and nature.
  Arms: Virtual Reality Glasses Group

SUMMARY:
The aim of the study was to examine the effects of the emotional freedom technique and virtual reality glasses applied to individuals receiving hyperbaric oxygen therapy for the first time on anxiety and vital signs. The hypotheses of this research are that there is a difference between the emotional liberation technique and virtual reality glasses groups and the control group in terms of anxiety and vital signs.

DETAILED DESCRIPTION:
This study was designed as a pretest-posttest regular parallel group, randomized controlled experimental. The research will be carried out in Konya City Hospital Hyperbaric Oxygen Therapy Unit. Patients will be randomly assigned to three groups: emotional freedom technique group (25), virtual reality glasses group (25) and control group (25). For Emotional Freedom Technique Group: The emotional freedom technique will be applied by the researcher who has received the practitioner training certificate. For Virtual Reality Glasses Group: The video containing the nature walk will be watched by virtual reality. For the Control Group: No intervention will be made in the control group. Standard care will be given. The primary result of this study is to determine the patients' anxiety scores. Secondary results of the research are to determine the patients' vital signs.

ELIGIBILITY:
İnclusion Criteria

* Applying HBO treatment for the first time,
* Volunteering to participate in the research,
* Those who are between the ages of 18 and 65,
* Able to speak and understand Turkish (patients who will not have communication problems),
* Without a psychiatric diagnosis,
* Those who have not received training on coping with anxiety and fear before,
* Those who have not attended a course on energy therapy before,
* Vital signs are within normal limits

Exclusion Criteria:

* Having hearing and vision problems,
* Urgently placed on HBO treatment,
* Patients without chronic diseases,
* Patients with impaired tissue integrity at EFT energy points

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 75 (Estimated)
Dates: Start 2024-10-01 (Estimated); Primary Completion 2024-10-01 (Estimated); Study Completion 2025-06-01 (Estimated)

PRIMARY OUTCOMES:
State Anxiety Inventory (STAI) | It will be applied within the first 10 minutes when the patient arrives at the Hyperbaric Oxygen treatment center, 10 minutes before the treatment and 10 minutes after the treatment.
  In the State Anxiety Inventory, the individual evaluates how he or she feels "at the moment" and according to the severity of the emotions or behaviors expressed in the items (1) "never", (2) "a little", (3) "a lot" and (4) "a lot".
  are asked to choose one of the statements "completely". The highest score of 4 is given for choosing the phrase "completely", and the lowest score is 1 for choosing the phrase "not at all". The lowest total score that can be obtained from the State Anxiety Scale is 20, and the highest total score is 80. A high score indicates a high level of anxiety, and a low score indicates a low level of anxiety.

SECONDARY OUTCOMES:
Blood Pressure | It will be applied within the first 10 minutes when the patient arrives at the Hyperbaric Oxygen treatment center, 10 minutes before the treatment and 10 minutes after the treatment.
  Blood pressure was evaluated with a sphygmomanometer. Accepted normal values: Systolic blood pressure: 100-120 mmHg, Diastolic blood pressure: 60-80 mmHg.
Pulse | It will be applied within the first 10 minutes when the patient arrives at the Hyperbaric Oxygen treatment center, 10 minutes before the treatment and 10 minutes after the treatment.
  Pulse was evaluated with a pulse oximeter device. Accepted normal values: 60-100 pulse /min
Respiration | It will be applied within the first 10 minutes when the patient arrives at the Hyperbaric Oxygen treatment center, 10 minutes before the treatment and 10 minutes after the treatment.
  Respiration was evaluated by observation. Accepted normal values:12-20 respiration /min
Body Temperature | It will be applied within the first 10 minutes when the patient arrives at the Hyperbaric Oxygen treatment center, 10 minutes before the treatment and 10 minutes after the treatment.
  It will be evaluated with a thermometer device. Accepted normal values: 36-37 ° C
Oxygen Saturation | It will be applied within the first 10 minutes when the patient arrives at the Hyperbaric Oxygen treatment center, 10 minutes before the treatment and 10 minutes after the treatment.
  Oxygen saturation was evaluated with a pulse oximetry device. Accepted normal values: SpO2: 95-100%.

CONTACTS AND LOCATIONS:
Overall Officials: gülsüm GÜRSOY AÇIKGÖZ, Principal Investigator — Necmettin Erbakan University
Locations (1):
- Gülsüm Gürsoy Açikgöz, Konya, Meram, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No